CLINICAL TRIAL: NCT07060040
Title: The Effects of a Dialysis-Specific Formula Rich in Branched-Chain Amino Acids, Omega-3, and Dietary Fiber on Nutritional Status
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Collaborators: Multipower Enterprise Corp. (Unknown)
Responsible Party: Principal Investigator, Yu-Li Lin, Director, Center for Chronic Kidney Disease Prevention and Care, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB114-018-A
Record Dates: First submitted 2025-06-20; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: ESRD (End-Stage Renal Disease); Dialysis
Keywords: Branched-chain amino acid; Protein-energy malnutrition; fiber; omega-3; oral nutritional supplements; dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Protein-Energy Malnutrition | interventions — Proteins; Fatty Acids, Omega-3; Dietary Fiber

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental formula (Experimental): BOSCOGEN 18% Protein ONS (240ml)
  Interventions: Dietary Supplement: BOSCOGEN 18% Protein ONS: Energy 480 kcal, Protein 21.6 g, BCAA 6000 mg, Omega-3 fatty acid 1.8 g, fiber 5 g
- comparative formula (Active Comparator): Fresubin dialysis ONS (200 ml)
  Interventions: Dietary Supplement: Fresubin dialysis ONS (200 ml): Energy 300 kcal, Protein 20 g, BCAA - mg, Omega-3 fatty acid - g, fiber 0.2 g

INTERVENTIONS:
Dietary Supplement: BOSCOGEN 18% Protein ONS: Energy 480 kcal, Protein 21.6 g, BCAA 6000 mg, Omega-3 fatty acid 1.8 g, fiber 5 g — Oral nutritional supplementation: Energy 480 kcal, Protein 21.6 g, BCAA 6000 mg, Omega-3 fatty acid 1.8 g, fiber 5 g
  Arms: Experimental formula
Dietary Supplement: Fresubin dialysis ONS (200 ml): Energy 300 kcal, Protein 20 g, BCAA - mg, Omega-3 fatty acid - g, fiber 0.2 g — Fresubin dialysis ONS (200 ml): Energy 300 kcal, Protein 20 g, BCAA - mg, Omega-3 fatty acid - g, fiber 0.2 g
  Arms: comparative formula

SUMMARY:
The aim of this study is to evaluate the effects of a specialized oral nutritional supplement (SF) enriched with BCAAs, omega-3 fatty acids, and dietary fiber on improving the nutritional status of dialysis patients with mild to moderate malnutrition, and thereby alleviating fatigue and enhancing quality of life. We will assess various aspects of protein-energy wasting (PEW), as well as changes in the Malnutrition Inflammation Score (MIS), Geriatric Nutritional Risk Index (GNRI), fatigue, appetite, serum BCAA levels, uremic toxins, and gut microbiota composition.

DETAILED DESCRIPTION:
Protein-energy wasting (PEW) is highly prevalent in dialysis patients. If not promptly addressed, PEW increases the risk of falls, disability, fractures, hospitalization, and mortality, while significantly impairing quality of life. In clinical care, nutritional supplementation can prevent the onset of PEW and improve quality of life by reducing the severity of malnutrition. Numerous studies and meta-analyses have shown that dietary fiber can help reduce uremic toxins in CKD and dialysis patients. Additionally, research has shown that the loss of branched-chain amino acids (BCAAs) during dialysis can lead to poor appetite, fatigue, and increased risk of PEW. In elderly hemodialysis patients, supplementation with 12 g/day of BCAAs has been shown to reduce anorexia and significantly improve nutritional status.

The aim of this study is to improve the nutritional status of dialysis patients with mild to moderate malnutrition by providing a specialized formula (SF) supplement enriched with branched-chain amino acids (BCAAs), omega-3 fatty acids, and dietary fiber. The ultimate goal is to alleviate fatigue and enhance quality of life. We will simultaneously evaluate changes in multiple aspects of protein-energy wasting (PEW), the malnutrition inflammation score (MIS), the Geriatric Nutritional Risk Index (GNRI), fatigue levels, appetite, serum BCAA concentrations, uremic toxins, and gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESRD who have been receiving dialysis for more than three months
* Serum albumin (Alb) ≤ 4.0 g/dL, or body mass index (BMI) ≤ 20, or normalized protein catabolic rate (nPCR) ≤ 0.8
* Male or female patients aged 20 years or older

Exclusion Criteria:

* Serum albumin (Alb) < 3.0 g/dL
* Known allergy or intolerance to any component of the product, or deemed by a physician to be unable to complete the trial
* Patients who refuse to sign the informed consent form or are unable to follow study instructions
* Pregnant or breastfeeding women
* Patients with severe illnesses (including burn injuries), undergoing major surgery, with abnormal liver function (GOT and GPT levels more than 5 times the upper limit of normal), or with malignancy (6) Participation in another clinical trial of investigational drugs or concurrent use of investigational drugs within 30 days prior to or during this trial (7) Any other serious medical condition as determined by the investigator that would make the patient unsuitable for participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Malnutrition Inflammation Score (MIS) | From enrollment to the end of treatment at 12 weeks
  Change in total score of MIS (range 0-30; higher scores indicate worse nutritional status)
Change in Geriatric Nutritional Risk Index (GNRI) | From enrollment to the end of treatment at 12 weeks
  Change in GNRI score calculated using serum albumin and body weight (higher scores indicate better nutritional status)
Change in serum albumin concentration | From enrollment to end of treatment (12 weeks)
  Change in serum albumin level (g/dL)
Change in serum pre-albumin concentration | From enrollment to end of treatment (12 weeks)
  Change in serum pre-albumin level (mg/dL)
Change in Protein-Energy Wasting (PEW) status | From enrollment to end of treatment (12 weeks)
  Change in PEW status based on ISRNM criteria (present/absent)
Change in body composition | From enrollment to end of treatment (12 weeks)
  Change in body composition including lean mass (kg) and fat mass (kg) as measured by bioimpedance

SECONDARY OUTCOMES:
Serum BCAA concentration | From enrollment to the end of treatment at 12 weeks
  Change in serum BCAA concentration
Serum indoxyl sulfate concentration | From enrollment to the end of treatment at 12 weeks
  Change in serum indoxyl sulfate level
Serum p-cresyl sulfate concentration | From enrollment to end of treatment (12 weeks)
  Change in serum p-cresyl sulfate level
Brief Fatigue Inventory - Taiwanese version | From enrollment to the end of treatment at 12 weeks
  Brief Fatigue Inventory - Taiwanese version (range 0-10; higher scores indicate greater fatigue)
Stool Form Assessment | From enrollment to the end of treatment at 12 weeks
  Bristol Stool Form Scale (a 7-point scale used to classify stool types, with higher score indicates looser stool consistency or more severe diarrhea)
Change in handgrip strength | From enrollment to end of treatment (12 weeks)
  Maximal and average handgrip strength (kg) will be measured using a hand dynamometer.

OTHER OUTCOMES:
Change in gut microbiota composition | From enrollment to the end of treatment at 12 weeks
  Gut microbiota composition (stool), Alpha and Beta diversity indices

IPD SHARING:
Plan to Share IPD: No